CLINICAL TRIAL: NCT02893748
Title: HyGIeaCare Prep vs Split-dose PEG Prep Prior to Colonoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to agree on budget terms
Sponsor: HyGIeaCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGP-0004
Record Dates: First submitted 2016-08-24; First posted 2016-09-08 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2018-02

CONDITIONS: Colonoscopy
Keywords: colon; polyps; cancer; screening
MeSH Terms: conditions — Polyps; Neoplasms | interventions — Colonoscopy; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1: HyGIeaCare Prep and Colonoscopy (Active Comparator): Patients will receive:
  1. HyGIeaCare Prep
  2. Colonoscopy
  Interventions: Device: HyGIeaCare Prep; Procedure: Colonoscopy
- 2: Split-dose PEG Prep and Colonoscopy (Active Comparator): Patients will receive:
  1. Split-dose PEG
  2. Colonoscopy
  Interventions: Procedure: Colonoscopy; Drug: polyethylene glycol (PEG)

INTERVENTIONS:
Device: HyGIeaCare Prep — Patients will receive the HyGIeaCare Prep, which is an open colon lavage system using warm water by gravity drip to evacuate the colon by stimulating peristalsis to cleanse the colon prior to colonoscopy.
  Other Names: colon lavage
  Arms: 1: HyGIeaCare Prep and Colonoscopy
Procedure: Colonoscopy — Screening colonoscopy as per standard of care.
  Other Names: Screening Colonoscopy
Drug: polyethylene glycol (PEG) — PEG preparation to be delivered in two doses - 1/2 the night before and 1/2 the morning of the colonoscopy
  Other Names: Split-dose PEG Prep
  Arms: 2: Split-dose PEG Prep and Colonoscopy

SUMMARY:
The purpose of this study is to compare the level of cleanliness using the HyGIeaCare Prep vs the standard of care Split-dose PEG prep used prior to colonoscopy.

DETAILED DESCRIPTION:
The level of cleanliness will be recorded using the Boston Bowel Prep Score (BBPS) by an endoscopist who is blind to the randomized preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred to colonoscopy
2. Patient with high probability for poor prep due to one or more of the following:

   1. Chronic constipation (Rome III functional constipation criteria)
   2. Gastroparesis
   3. Immobilization
   4. Diabetes
   5. History of poor prep

Exclusion Criteria:

1. Patient has any condition that, in the opinion of the investigator, may adversely affect the compliance or safety of the patient or would limit the patient's ability to complete the study.
2. Patient is currently taking narcotics.
3. Patient has any of the contraindications listed below:

   1. Cardiac: Congestive heart failure (NYHA class III or IV or EF < 50%)
   2. GI: Intestinal perforation, carcinoma of the rectum, fissures or fistula, severe hemorrhoids, abdominal hernia, recent colon or rectal surgery, or abdominal surgery
   3. GU: Renal insufficiency (CC < 60 ml/min/173m2), cirrhosis with ascites
   4. Abdominal surgery within the last 6 months
   5. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Colon cleanliness will be measured in both groups according to the Boston Bowel Preparation Scale (BBPS) | Day 1 of colonoscopy

SECONDARY OUTCOMES:
Evaluation of patient satisfaction using a Questionnaire | 2 Days after colonoscopy
  Questionnaire
Evaluation of adverse events | 2 Days after colonoscopy
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Umar, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK; US Multi-Society Task Force on Colorectal Cancer. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the US multi-society task force on colorectal cancer. Gastroenterology. 2014 Oct;147(4):903-24. doi: 10.1053/j.gastro.2014.07.002. No abstract available. PMID 25239068
- [Background] Gagneja HK, Parekh P, Burleson D, Johnson D. HyGIeaCare® Preparation for Colonoscopy - A Technical Update for Success. J Gastrointest Dig Syst 2016; 6: 458. doi:10.4172/2161-069X.1000458
- [Background] Clark BT, Protiva P, Nagar A, Imaeda A, Ciarleglio MM, Deng Y, Laine L. Quantification of Adequate Bowel Preparation for Screening or Surveillance Colonoscopy in Men. Gastroenterology. 2016 Feb;150(2):396-405; quiz e14-5. doi: 10.1053/j.gastro.2015.09.041. Epub 2015 Oct 9. PMID 26439436
- [Background] Fiorito J, Culpepper-Morgan JA, Estabrook SG, Scofield P, Usatii V, Cuomo R. Hydrotherapy Compared with PEG-ES Lavage and Aqueous Sodium Phosphate as Bowel Preparation for Elective Colonoscopy: A Prospective, Randomized, Single Blinded Trial. ACG Abstract 2006; 751814.
- [Background] Sportes A, Delvaux M, Huppertz J, Hernandez C, Gay G. Randomized Trial Comparing High Volume Rectal Water Irrigation with Standard 4L Split-dose PEG Preparation Before Colonoscopy. Accepted by Gastroenterology and Digestive Diseases (awaiting publication).
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062
- [Background] US Department of Health and Human Services. Common Terminology Criteria for Adverse Events 2009.